CLINICAL TRIAL: NCT01551953
Title: BEAM COPD: Breathing, Education, Awareness and Movement in Chronic Obstructive Pulmonary Disease
Brief Title: BEAM COPD: Breathing, Education, Awareness and Movement in Chronic Obstructive Pulmonary Disease (COPD)
Acronym: BEAM COPD
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Beth Israel Deaconess Medical Center (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Center for Complementary and Integrative Health (NCCIH) (NIH)
Responsible Party: Principal Investigator, Gloria Y. Yeh, Associate Professor of Medicine, Beth Israel Deaconess Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 2010P000412; R01AT005436 (NIH)
Record Dates: First submitted 2012-03-01; First posted 2012-03-13 (Estimated); Last update posted 2017-02-27 (Actual); Status verified 2017-02

CONDITIONS: Chronic Obstructive Pulmonary Disease (COPD)
Keywords: chronic bronchitis; emphysema; pulmonary; COPD
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Bronchitis, Chronic; Emphysema | interventions — Tai Ji; Educational Status

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- tai chi exercise (Experimental)
  Interventions: Behavioral: Tai chi
- mind-body breathing (Experimental)
  Interventions: Behavioral: Mind-body breathing
- education (Active Comparator)
  Interventions: Behavioral: Education

INTERVENTIONS:
Behavioral: Tai chi — 12 week tai chi class
  Arms: tai chi exercise
Behavioral: Mind-body breathing — 12 week breathing class
  Arms: mind-body breathing
Behavioral: Education — 12 week education class
  Arms: education

SUMMARY:
The main purpose of this study is to determine feasibility and effects of tai chi and mind-body breathing in patients with COPD.

ELIGIBILITY:
Inclusion Criteria:

1. Moderate-severe COPD
2. Age ≥ 40 years

Exclusion Criteria:

1. Subjects with respiratory failure or GOLD stage 4 who are unable to safely perform a 6 minute walk test or otherwise safely exercise as deemed by a physician.
2. COPD exacerbation requiring steroids, antibiotics, ED visit or hospitalization within the past 2 weeks unless physician deems subject at baseline
3. Planned major pulmonary intervention within the next 3 months
4. Hypoxemia on walk test or cardiopulmonary exercise test
5. Inability to ambulate due to vascular or other neuromuscular conditions that would preclude a walk test
6. Clinical signs of unstable cardiovascular disease
7. Severe cognitive dysfunction
8. Non-English speaking
9. Current active participation in pulmonary rehabilitation program or current regular practice of tai chi
10. Physician diagnosis of unstable/untreated clinical depression
11. History of lung cancer

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 124 (Actual)
Dates: Start 2011-02; Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Feasibility of tai chi intervention | 12 weeks
  Willingness to participate, adherence, and safety

SECONDARY OUTCOMES:
Change from baseline- Disease specific quality of life | baseline, 12 weeks, 24 weeks
  Chronic Respiratory Questionnaire
Change from baseline- Exercise capacity | baseline, 12 weeks, 24 weeks
  six-minute walk distance, cardiopulmonary exercise testing
Change from baseline- Dyspnea | baseline, 12 weeks, 24 weeks
  UCSD Shortness of Breath Questionnaire
Change from baseline- Psychosocial well-being | baseline, 12 weeks, 24 weeks
  CES-D, Perceive Stress Scale, COPD Self-Efficacy Scale, Multidimensional Scale of Percieved Social Support
Change from baseline- Pulmonary function | baseline, 12 weeks, 24 weeks
  Spirometry and lung volumes
Change from baseline- Physical strength and flexibility | baseline, 12 weeks, 24 weeks
  Chair Sit and Reach, Chair Stand

CONTACTS AND LOCATIONS:
Overall Officials: Gloria Yeh, MD, MPH, Principal Investigator — BIDMC, Harvard Medical School
Locations (2):
- United States (2):
  - VA Healthcare System, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts

REFERENCES:
- [Derived] Kraemer KM, Kilgore K, Litrownik D, Jean-Laurent B, Wayne PM, Richardson CR, Moy ML, Yeh GY. A Web-Based Mind-Body Intervention (Mindful Steps) for Promoting Walking in Chronic Cardiopulmonary Disease: Insights From a Qualitative Study. Glob Adv Integr Med Health. 2023 Dec 2;12:27536130231212169. doi: 10.1177/27536130231212169. eCollection 2023 Jan-Dec. PMID 38050584
- [Derived] Gilliam EA, Cheung T, Kraemer K, Litrownik D, Wayne PM, Moy ML, Yeh GY. The impact of Tai Chi and mind-body breathing in COPD: Insights from a qualitative sub-study of a randomized controlled trial. PLoS One. 2021 Apr 8;16(4):e0249263. doi: 10.1371/journal.pone.0249263. eCollection 2021. PMID 33831022
- [Derived] Yeh GY, Litrownik D, Wayne PM, Beach D, Klings ES, Reyes Nieva H, Pinheiro A, Davis RB, Moy ML. BEAM study (Breathing, Education, Awareness, Movement): a randomised controlled feasibility trial of tai chi exercise in patients with COPD. BMJ Open Respir Res. 2020 Nov;7(1):e000697. doi: 10.1136/bmjresp-2020-000697. PMID 33219007
- [Derived] Yeh GY, Wayne PM, Litrownik D, Roberts DH, Davis RB, Moy ML. Tai chi mind-body exercise in patients with COPD: study protocol for a randomized controlled trial. Trials. 2014 Aug 28;15:337. doi: 10.1186/1745-6215-15-337. PMID 25168853